CLINICAL TRIAL: NCT05786651
Title: Task Switching Behavior Between Target Templates During Visual Search in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lehigh University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 6R15EY030247-01A1 (NIH)
Record Dates: First submitted 2023-03-15; First posted 2023-03-27 (Actual); Results first posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Healthy
Keywords: attention; visual search

STUDY DESIGN:
Intervention Model Description: All participants receive each level of visual information (target or distractor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Within-Subjects Attentional Information (Experimental): Within-Subjects, all participants receive all interventions
  Interventions: Behavioral: Experimental: Within-Subjects Attentional Information

INTERVENTIONS:
Behavioral: Experimental: Within-Subjects Attentional Information — Visual Search Information Type (target or distractor information) Participants will have information about targets, distractors, or neither in different trials of the intervention.

SUMMARY:
In this line of research, the researchers having participants engage in task switching between tasks which require a positive (target) template, negative (distractor) template, or neutral (non-informative) template to the cognitive control factors associated with each template type during visual search. This is a basic science study.

DETAILED DESCRIPTION:
The researchers will have participants engage in task switching between tasks which require a positive (target) template, negative (distractor) template, or neutral (non-informative) template to the cognitive control factors associated with each template type during visual search. Looking for impacts of task switching helps to identify the components of the cognitive control system that overlap between different types of attentional templates. This is a basic science study.

ELIGIBILITY:
Inclusion Criteria:

* normal or corrected to normal visual acuity, normal color vision

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-10-17 (Actual); Primary Completion 2018-11-09 (Actual); Study Completion 2018-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Carlisle, Principal Investigator — Lehigh University
Locations (1):
- Lehigh University, Bethlehem, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The researchers plan to share anonymized subject data on Open Science Framework.
Supporting Information: Study Protocol, SAP
Time Frame: Upon publication.
Access Criteria: Open Science Framework internet access.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Lehigh University, normal or corrected to normal visual acuity and normal color vision
Period: Overall Study
Arm/Group | Within-Subjects Attentional Information
Started | 27
Completed | 26
Not Completed | 1
Not completed — fire alarm during testing session, incomplete testing | 1

BASELINE CHARACTERISTICS:
Arm/Group | Within-Subjects Attentional Information
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.07 (1.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Button Press Reaction Time
Description: Speed to respond correctly to the target- after participant finds the target shape on a computer screen, they press a button to indicate what shape they see
Time Frame: One day (during testing)
Population: Two participants were removed due to low accuracy (2 standard deviations below the mean) in one or more conditions.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Within-Subjects Attentional Information
Number analyzed (Participants) | 24
Seconds
  Positive cue: repeat cue meaning, repeat cue color | 1.68 (.03)
  Positive cue: repeat cue meaning, change cue color | 1.69 (.03)
  Positive cue: Change Meaning, repeat color | 1.76 (.04)
  Positive cue: cue meaning change, cue color change | 1.77 (.04)
  Negative cue: repeat cue meaning, repeat cue color | 1.93 (.03)
  Negative cue: repeat cue meaning, change cue color | 1.97 (.03)
  Negative cue: Change Meaning, repeat color | 1.78 (.03)
  Negative cue: cue meaning change, cue color change | 1.88 (.03)
Statistical Analysis 1: Comparison: Within-Subjects Attentional Information; Test type: Equivalence — Comparison of conditions; p < .05, ANOVA

2. Primary Outcome: Button Press Accuracy
Description: Accuracy of responses to target item (% correct)- the researchers will measure whether the participants presses the correct button which corresponds to the target shape presented on the computer screen or the incorrect button
Time Frame: One day (during testing)
Population: Two participants were removed due to low accuracy (2 standard deviations below the mean) in one or more conditions.
Measure: Mean (Standard Error); unit: proportion correct
Arm/Group | Within-Subjects Attentional Information
Number analyzed (Participants) | 24
proportion correct
  Positive cue: repeat cue meaning, repeat cue color | .912 (.008)
  Positive cue: repeat cue meaning, change cue color | .926 (.017)
  Positive cue: Change Meaning, repeat color | .875 (.014)
  Positive cue: cue meaning change, cue color change | .852 (.014)
  Negative cue: repeat cue meaning, repeat cue color | .843 (.017)
  Negative cue: repeat cue meaning, change cue color | .819 (.022)
  Negative cue: Change Meaning, repeat color | .873 (.016)
  Negative cue: cue meaning change, cue color change | .835 (.016)
Statistical Analysis 1: Comparison: Within-Subjects Attentional Information; Test type: Equivalence — Comparisons of mean values of conditions; p < .05, ANOVA

ADVERSE EVENTS:
Time Frame: Day of testing
Description: This study is a simple behavioral intervention, examining performance on a computer-based cognitive psychology task. There were no expected risks beyond typical daily computer use, which may include headache from looking at at a computer screen or boredom. No serious adverse events were expected. Research assistants monitored for unanticipated adverse effects.
Arm/Group | Within-Subjects Attentional Information
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-10): https://cdn.clinicaltrials.gov/large-docs/51/NCT05786651/Prot_SAP_000.pdf